CLINICAL TRIAL: NCT02520193
Title: Prospective, Randomized, Multi-center Trial to Assess the Impact of Early Mobilization on Mechanical Ventilation Duration in Intubated Critically Ill Patients
Brief Title: Impact of Early Mobilization on Mechanical Ventilation Duration in Intubated Critically Ill Patients
Acronym: EarlyMob
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHRIP 2014-01; 2015-A00741-48 (Other: ANSM)
Record Dates: First submitted 2015-07-28; First posted 2015-08-11 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2016-07

CONDITIONS: ICU Acquired Weakness
Keywords: Early mobilisation; Invasive ventilation; Ventilator free days; Intensive Care Unit
MeSH Terms: interventions — Intensive Care Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard mobilization strategy (No Intervention)
- protocolized early mobilization strategy (Experimental)
  Interventions: Procedure: Protocolized early mobilization in ICU

INTERVENTIONS:
Procedure: Protocolized early mobilization in ICU
  Arms: protocolized early mobilization strategy

SUMMARY:
The purpose of the present study is to compare usual care in terms of mobilization performed to intubated ICU patients to a standardized program designed to deliver early mobilization at least 5 days a week.

This study has a before / after design with a control group during the experimental phase. The first phase of the study corresponds to an observational phase during which every act of mobilization performed to the included patients is going to be documented. During this first study period, total duration of mechanical ventilation is going to be recorded for all the patients included.

At the end of this first study period, the participating ICU are going to be randomized (Cluster randomization) in two groups either observational or experimental. The corresponding strategy is going to be applied to all the patients included during the second study period. During this second period, total duration of mechanical ventilation is also going to be recorded for all the patients included.

The study hypothesis is that applying a protocolized early mobilization strategy increases the number of ventilator free-days during the 28 days after intubation in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission in intensive care unit
* Invasive ventilation for more than 24 hours
* Invasive ventilation for less than 48 hours
* Expected duration of invasive ventilation of more than 24 hours at the time of inclusion.

Exclusion Criteria:

* Pregnancy
* Failure to obtain a consent from someone authorized
* Patient under law protection.
* Patient non-affiliated to a health care system.
* Active therapeutic limitation
* Hospitalisation for more than 7 days before intubation
* Admission in intensive care unit after a surgical procedure, burn or trauma
* Admission in intensive care unit because of neurological disease
* Previously known neuromuscular disease
* Bilateral lower limbs amputation
* BMI above 40 kg/m²
* Limitation in daily activities before ICU admission
* Chronic ventilation (more than 12h /24 hours) on tracheotomy before ICU admission
* Participation in another interventional clinical study related to mobilization or in an interventional clinical study which has mechanical ventilation duration as primary outcome
* Previous enrolment in the same phase of the EarlyMob study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Number of days without mechanical ventilation (ventilator-free days) during the 28 days after intubation | 28 days after intubation

SECONDARY OUTCOMES:
The incidence of Intensive Care Unit-acquired weakness with Manual Muscle Testing (MMT) scale | end of Intensive Care Unit stay, an expected average of 10 days
The incidence and stage of pressure ulcers occurring during ICU stay with NPUAP scale | end of Intensive Care Unit stay, an expected average of 10 days
The incidence of delirium with CAM-ICU scale | end of Intensive Care Unit stay, an expected average of 10 days
Hospital stay duration | End of hospital stay, an expected average of 20 days
Place where the patient is transferred at the end of the hospital stay | End of hospital stay, an expected average of 20 days
The delay, in number of days between intubation and the first successful spontaneous breathing trial | End of Intensive Care Unit stay, an expected average of 10 days
The incidence of extubation failure defined as re-intubation within 72 hours after the first extubation | end of Intensive Care Unit stay, an expected average of 10 days
Time between intubation and the first stand-up position in days | end of Intensive Care Unit stay, an expected average of 10 days
ICU stay duration | end of Intensive Care Unit stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Locations (23):
- Belgium (5):
  - Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc - Service des soins intensifs, Brussels
  - CHR Citadelle - Services Soins intensifs, gériatriques et pédiatriques, Liège
  - CHU de Liege - Service de soins intensifs généraux, Liège
  - Cliniques Universitaires UCL de Mont-Godinne - Service intensifs généraux, Yvoir
- France (17):
  - CHU Angers - Service de Réanimation Médicale et de Médecine Hyperbare, Angers
  - CHU de Brest - Service de réanimation médicale, Brest
  - CH de Pontoise - Serive de réanimation médicale - CH René Dubos, Cergy-Pontoise
  - AP-HP Hôpital Henri Mondor - Service de Réanimation Médicale, Créteil
  - CHD Vendée - Service de Réanimation Polyvalente, La Roche-sur-Yon
  - Centre Hospitalier La Rochelle - Ré- Aunis - Réanimation polyvalente, La Rochelle
  - CHU Grenoble - Service de Réanimation Médicale - Hôpital A, Michallon, La Tronche
  - Centre Hospitalier Le Mans - Service de Réanimation médico-chirurgicale, Le Mans
  - CHRU de Lille - Pôle de réanimation -Hôpital Roger Salengro, Lille
  - CH St Joseph St Luc - Service de Réanimation Polyvalente, Lyon
  - Groupe Hospitalier du Havre - Service de Réanimation médico-chirurgicale - Hôpital Jacques Monod, Montivilliers
  - CHU de Nantes - Service de Réanimation Médicale Polyvalente, Nantes
  - CHU de Nice - Service de réanimation médicale - Hôpital de l'Archet, Nice
  - AP-HP Hôpital Tenon - Service de Réanimation, Paris
  - AP-HP Hôpitaux Universitaires Paris Ouest- Service de réanimation médicale - Hôpital Européen Georges Pompidou, Paris
  - CHU Toulouse - service de néphrologie Hémodialyse HTA Transplantation d'Organes - Hôpital Rangueil, Toulouse
  - Service de Réanimation Polyvalente -CHU de Toulouse - Hôpital Rangueil, Toulouse
- CHUV, Lausanne, Switzerland